CLINICAL TRIAL: NCT01422837
Title: VIvitrol's Cost and Treatment Outcomes RegistrY
Brief Title: ALK21-025: Vivitrol's Cost and Treatment Outcomes Registry
Acronym: VICTORY
Status: Completed | Type: Observational
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALK21-025
Record Dates: First submitted 2011-08-23; First posted 2011-08-24 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Opioid Dependence
Keywords: opioid; dependence; VIVITROL
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the VIVITROL Registry is to gather real world data on opioid dependence and to provide understanding of the health economics of opioid dependence.

DETAILED DESCRIPTION:
The VIVITROL Registry is an observational, open-label, single-arm, multi-center registry of patients who have initiated treatment with VIVITROL for prevention of relapse to opioid dependence, following opioid detoxification.

The objectives of the VIVITROL Registry are:

* To describe characteristics of patients receiving VIVITROL for opioid dependence in real-world clinical practice.
* To assess clinical, health economic, and health-related quality of life (HRQOL) outcomes in a broad population of patients receiving VIVITROL in real-world clinical practice.
* To provide additional data to inform future research on VIVITROL.

Patients 18 years of age or older who have been determined by their participating prescriber to be an appropriate candidate for VIVITROL treatment may be offered enrollment into the registry. The decision to treat a patient with VIVITROL will be made by the patient's participating prescriber independent of the registry. VIVITROL will not be provided to patients enrolled in the registry in exchange for their participation; patients will receive commercially available VIVITROL via a standard prescription that will be filled through standard commercial channels.

Patients will be observed while receiving VIVITROL and for six months after they discontinue VIVITROL use. The registry is non-interventional; it will neither direct the treatment plan for enrolled patients nor define the frequency of follow-up visits of each patient. A patient's participation in the registry will not influence or direct patient treatment procedures or follow-up care. It is expected that patients will be seen at least once per month during active VIVITROL treatment to receive their monthly injection.

During the standard monthly injection visits, patients will be asked to provide detailed health economics information using a variety of questionnaires, including the EQ-5D and SF-12v2.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 18 years or older
* Patient is diagnosed with a current opioid dependence for which treatment with VIVITROL is being initiated
* Patient has provided written informed consent
* Patient is willing and able to provide the information to be collected via the registry's interviews and questionnaires
* Patient expects to be available for ongoing registry participation

Exclusion Criteria:

* Prior use of VIVITROL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The VIVITROL Registry will enroll patients who have been prescribed VIVITROL for the prevention of relapse to opioid dependence, following opioid detoxification.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (31):
- United States (31):
  - Assisted Recovery Centers of America, Phoenix, Arizona
  - Arkansas Psychiatric Clinc, Little Rock, Arkansas
  - Amy Solomon, MD, Ben Lomond, California
  - Touchstone Medical Group, Clovis, California
  - Kenneth C. Russ, MD, Palm Springs, California
  - Tarzana Treatment Centers, Tarzana, California
  - The NeuroBehavioral Institute of Colorado, PC, Lone Tree, Colorado
  - Psychotherapy Services, Etc., Groton, Connecticut
  - Jacqueline Boutrouille, MD, Tamarac, Florida
  - Alliance Clinical Research, Winter Park, Florida
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - PACT Atlanta, Decatur, Georgia
  - Gosnold-Thorne Counseling Center, Centerville, Massachusetts
  - Dr. Li's Clinic, Milford, Massachusetts
  - Assisted Recovery Centers of America, St Louis, Missouri
  - Dent Neurologic Institute, Amherst, New York
  - Dr. Michael Sanders, Great Neck, New York
  - Fakhouri Medical, Hopewell Junction, New York
  - Parallax Center, New York, New York
  - Healing Comfort Clinic, Corvallis, Oregon
  - Jasper Health, Media, Pennsylvania
  - Institute of Addiction Medicine, Plymouth Meeting, Pennsylvania
  - Innovation Laboratory/PEARL, Johnson City, Tennessee
  - Urschel Recovery Science Institute, Dallas, Texas
  - Holiner Psychiatric Group, Dallas, Texas
  - Lenae White, MD, PA, Dallas, Texas
  - Utah Addiction Medicine & Counseling, Bountiful, Utah
  - Adolescent and Family Health Center, PC, Midlothian, Virginia
  - Chessen and Associates, Newport News, Virginia
  - Creekside Center for Integrative Medicine, Bellevue, Washington
  - Child and Adolescent Psychiatry, Bothell, Washington

REFERENCES:
- [Result] Saxon AJ, Akerman SC, Liu CC, Sullivan MA, Silverman BL, Vocci FJ. Extended-release naltrexone (XR-NTX) for opioid use disorder in clinical practice: Vivitrol's Cost and Treatment Outcomes Registry. Addiction. 2018 Aug;113(8):1477-1487. doi: 10.1111/add.14199. Epub 2018 Apr 1. PMID 29493836